CLINICAL TRIAL: NCT02637115
Title: Evaluation of the Effects Associated With the Administration of Akkermansia Muciniphila on Parameters of Metabolic Syndrome Related to Obesity
Brief Title: Evaluation of the Effects Associated With the Administration of Akkermansia Muciniphila on Parameters of Metabolic Syndrome
Acronym: Microbes4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrice D. Cani (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor-Investigator, Patrice D. Cani, Professor, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015/02JUL/369; B403201525111 (Other: Université catholique de Louvain)
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Syndrome x; Glucose Metabolism Disorders; Dyslipidemias; Obesity
Keywords: Gut microbiota; Akkermansia muciniphila
MeSH Terms: conditions — Metabolic Syndrome; Glucose Metabolism Disorders; Dyslipidemias; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Subjects and physicians were both blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo corresponds to a solution of Phosphate buffer saline (PBS) and glycerol, that is the carrier used in the 3 other groups receiving the bacteria (active arms)
  Interventions: Dietary Supplement: Placebo
- Live Akk 9 (Experimental): Live Akkermansia muciniphila (Akk) at the dose of 10exp9 live bacteria (one billion of live bacteria) per day
  Interventions: Dietary Supplement: Live Akk 9
- Live Akk 10 (Experimental): Live Akkermansia muciniphila (Akk) at the dose of 10exp10 live bacteria (ten billion of live bacteria) per day
  Interventions: Dietary Supplement: Live Akk 10
- Killed Akk (Experimental): This group corresponds to Akkermansia muciniphila that have been heat-killed. The initial quantity of bacteria before the heating procedure was of 10exp10 bacteria.
  Interventions: Dietary Supplement: Killed Akk

INTERVENTIONS:
Dietary Supplement: Placebo — Consumption of one dose-sachet per day. This dose-sachet contains a placebo (PBS/Glycerol)
  Arms: Placebo
Dietary Supplement: Live Akk 9 — Consumption of one dose-sachet per day. This dose-sachet contains Live Akkermansia muciniphila (one billion per dose-sachet)
  Arms: Live Akk 9
Dietary Supplement: Live Akk 10 — Consumption of one dose-sachet per day. This dose-sachet contains Live Akkermansia muciniphila (ten billion per dose-sachet)
  Arms: Live Akk 10
Dietary Supplement: Killed Akk — Consumption of one dose-sachet per day. This dose-sachet contains heat-killed Akkermansia muciniphila
  Arms: Killed Akk

SUMMARY:
Overweight and obesity have reached worldwide epidemic level. Both overweight and obesity are characterized by comorbidities such as cardio-metabolic risk factors (i.e., insulin resistance, type 2 diabetes, hypertension, dyslipidemia, low-grade inflammation) representing a major public health problem. Therefore, it is urgent to find a therapeutic solution to target all these metabolic disorders. Among the environmental factors able to influence the individual susceptibility to gain weight and to develop metabolic disorders associated with obesity, more and more evidence show that the trillions of bacteria housed in our gastro-intestinal tract (i.e, gut microbiota) influence host metabolism. The investigators recently discovered a putative interesting microbial candidate, namely Akkermansia muciniphila (Akk). More exactly, we found that the administration of Akkermansia muciniphila reduced body weight gain, fat mass gain, glycemia and inflammatory markers in diet-induced obese mice. Moreover, in overweight/obese patients with cardiovascular risk factors subjected to a calorie restriction diet (calorie restriction diet for 6 weeks and an additional 6 weeks of weight maintenance), a higher abundance of Akkermansia muciniphila was associated with a better cardio-metabolic status in these patients. The investigators also discovered that patients having more Akkermansia muciniphila in their gut before the calorie restriction exhibited a greater improvement in glucose homoeostasis, blood lipids and body composition after calorie restriction. These observations suggested that the administration of Akkermansia muciniphila in overweight or obese people could be a very interesting therapeutic solution. Currently, no human study has investigated the beneficial effects of Akkermansia muciniphila administration on obesity and metabolic disorders. The overall objective of this study is to evaluate the effects associated with the administration of live or heat-killed Akkermansia muciniphila on the metabolic disorders (insulin-resistance, type-2 diabetes, dyslipidemia, inflammation) related to overweight and obesity in humans.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old
* Caucasian
* Insulin resistance (based on HOMA single-value)
* BMI between 25 and 50 kg/m²
* Metabolic syndrome: presence of at least 3 of the following criteria

  * Hypertension (blood pressure ≥ 130/85 mm Hg or antihypertensive treatment)
  * Hypertriglyceridemia (triglyceridemia ≥ 150mg/dl)
  * Low HDL-cholesterol (HDL-cholesterol < 40mg/dl for males, 50mg/dl for females)
  * Visceral obesity (waist circumference > 102 cm for males, 88cm for females)
  * Fasting hyperglycemia (fasting glycemia ≥ 110mg/dl)
* Informed consent signed by the patient

Exclusion Criteria:

* Acute or chronic progressive or chronic unstabilized diseases
* Alcohol consumption (more than 2 glasses per day)
* Previous bariatric surgery
* Surgery in the 3 months prior the study or surgery planned in the next 6 months
* Pregnancy or pregnancy planned in the next 6 months
* More than 30 minutes of sports 3 times per week
* Consumption of dietary supplement (omega-3 fatty acids, probiotics, prebiotics, plant stanols/sterols) in the month prior the study
* Inflammatory bowel disease or irritable bowel syndrome
* Diabetic gastrointestinal autonomic neuropathy (such as gastroparesis or reduced gastrointestinal motility)
* Consumption of more than 30g of dietary fibers per day
* Vegetarian or unusual diet
* Lactose intolerance or milk protein allergy
* Gluten intolerance
* Medications influencing parameters of interest (antidiabetic drugs such as metformin, DPP-4 inhibitors, GLP-1 receptor agonists, acarbose, hypoglycemic sulfonamides,glinides, thiazolidinediones, SGLT2 inhibitors, insulin,lactulose, consumption of antibiotics in the 2 months prior the study, corticosteroids, immunosuppressive agents, statins, fibrate, orlistat, cholestyramine, ezetimibe)
* Glycated hemoglobin (HbA1c) > 7.5%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Tolerance | 15 days
  self reporting of gastrointestinal symptoms (nausea, bloating, flatulence, cramp, borborygmi and gastric reflux)
Tolerance | 3 months
  self reporting of gastrointestinal symptoms (nausea, bloating, flatulence, cramp, borborygmi and gastric reflux)
Concentration of urea (mg/dl) | 15 days
  measure of urea as marker of renal function
Concentration of urea (mg/dl) | 3 months
  measure of urea as marker of renal function
Glomerular filtration rate (mL/min/1.73m2) | 15 days
  measure of glomerular filtration rate as marker of renal function
Glomerular filtration rate (mL/min/1.73m2) | 3 months
  measure of glomerular filtration rate as marker of renal function
Concentration of creatinine (mg/dl) | 15 days
  measure of creatinine as marker of renal function
Concentration of creatinine (mg/dl) | 3 months
  measure of creatinine as marker of renal function
Concentration of liver transaminases | 15 days
  measure of alanine aminotransferase (U/L); aspartate aminotransferase (U/L); gamma glutamyl transpeptidase (U/L). Lactate dehydrogenase (UI/L) as markers of hepatic inflammation
Concentration of liver transaminases | 3 months
  measure of alanine aminotransferase (U/L); aspartate aminotransferase (U/L); gamma glutamyl transpeptidase (U/L). Lactate dehydrogenase (UI/L) as markers of hepatic inflammation
Concentration of white blood cells (10exp3/µl) | 15 days
  measured as a marker of inflammation
Concentration of white blood cells (10exp3/µl) | 3 months
  measured as a marker of inflammation
concentration of CRP (c-reactive protein) (mg/dl) | 15 days
  measured as a marker of inflammation
concentration of CRP (c-reactive protein) (mg/dl) | 3 months
  measured as a marker of inflammation
Insulin resistance | 3 months
  HOMA-Homeostasis Model Assessment calculated from fasted glycemia and insulinemia
Concentration of blood lipids | 3 months
  Analysis of circulating lipids : total, LDL and HDL cholesterol (mg/dl), triglycerides (md/dl)
Obesity | 3 months
  Body weight
Adiposity | 3 months
  Fat mass evaluated by bioimpedance measurements
Visceral adiposity | 3 months
  Waist and hip circumference

SECONDARY OUTCOMES:
Measure of the concentration of Akkermansia in the feces (bacterial cells/g of feces) | 3 months
  Metagenomic analysis of the gut bacteria by using sequencing technology and by using quantitative polymerase chain reaction (qPCR).
Gut barrier function | 3 months
  Fecal calprotectin, fecal zonulin, plasma lipopolysaccharides (LPS) binding protein (LBP)
Metabolic endotoxemia | 3 months
  Plasma lipopolysaccharides (LPS) by the limulus amebocyte lysate kinetic chromogenic methodology
Gut microbial-related metabolites in urine | 3 months
  Metabolomic analysis of the bacterial metabolites present in the urine by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry
Gut microbial-related metabolites in plasma | 3 months
  Metabolomic analysis of the bacterial metabolites present in the plasma by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Patrice D. Cani, Professor, Study Director — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schneeberger M, Everard A, Gomez-Valades AG, Matamoros S, Ramirez S, Delzenne NM, Gomis R, Claret M, Cani PD. Akkermansia muciniphila inversely correlates with the onset of inflammation, altered adipose tissue metabolism and metabolic disorders during obesity in mice. Sci Rep. 2015 Nov 13;5:16643. doi: 10.1038/srep16643. PMID 26563823
- [Background] Dao MC, Everard A, Aron-Wisnewsky J, Sokolovska N, Prifti E, Verger EO, Kayser BD, Levenez F, Chilloux J, Hoyles L; MICRO-Obes Consortium; Dumas ME, Rizkalla SW, Dore J, Cani PD, Clement K. Akkermansia muciniphila and improved metabolic health during a dietary intervention in obesity: relationship with gut microbiome richness and ecology. Gut. 2016 Mar;65(3):426-36. doi: 10.1136/gutjnl-2014-308778. Epub 2015 Jun 22. PMID 26100928
- [Background] Everard A, Belzer C, Geurts L, Ouwerkerk JP, Druart C, Bindels LB, Guiot Y, Derrien M, Muccioli GG, Delzenne NM, de Vos WM, Cani PD. Cross-talk between Akkermansia muciniphila and intestinal epithelium controls diet-induced obesity. Proc Natl Acad Sci U S A. 2013 May 28;110(22):9066-71. doi: 10.1073/pnas.1219451110. Epub 2013 May 13. PMID 23671105
- [Derived] Depommier C, Vitale RM, Iannotti FA, Silvestri C, Flamand N, Druart C, Everard A, Pelicaen R, Maiter D, Thissen JP, Loumaye A, Hermans MP, Delzenne NM, de Vos WM, Di Marzo V, Cani PD. Beneficial Effects of Akkermansia muciniphila Are Not Associated with Major Changes in the Circulating Endocannabinoidome but Linked to Higher Mono-Palmitoyl-Glycerol Levels as New PPARalpha Agonists. Cells. 2021 Jan 19;10(1):185. doi: 10.3390/cells10010185. PMID 33477821
- [Derived] Depommier C, Flamand N, Pelicaen R, Maiter D, Thissen JP, Loumaye A, Hermans MP, Everard A, Delzenne NM, Di Marzo V, Cani PD. Linking the Endocannabinoidome with Specific Metabolic Parameters in an Overweight and Insulin-Resistant Population: From Multivariate Exploratory Analysis to Univariate Analysis and Construction of Predictive Models. Cells. 2021 Jan 5;10(1):71. doi: 10.3390/cells10010071. PMID 33466285